CLINICAL TRIAL: NCT05118776
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Multi-center Trial to Evaluate Safety and Efficacy pf ASC40 Tablets Combined With Bevacizumab in Subjects With Recurrent Glioblastoma
Brief Title: Study to Evaluate the Safety and Efficacy of ASC40 Tablets in Combination With Bevacizumab in Subjects With rGBM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC40-301
Record Dates: First submitted 2021-10-26; First posted 2021-11-12 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Recurrent Glioblastoma
Keywords: ASC40; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — TVB-2640; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASC40 (Experimental): ASC40 tablets 100mg/m^2 and bevacizumab 10mg/kg.
  Interventions: Drug: ASC40 tablets; Drug: Bevacizumab
- Placebo (Placebo Comparator): Placebo and bevacizumab 10mg/kg.
  Interventions: Drug: Placebo tablets; Drug: Bevacizumab

INTERVENTIONS:
Drug: ASC40 tablets — ASC40 tablets administered orally once daily
  Other Names: TVB-2640
  Arms: ASC40
Drug: Placebo tablets — Placebo administered orally once daily.
  Arms: Placebo
Drug: Bevacizumab — Bevacizumab once every 2 weeks, intravenous drip.

SUMMARY:
This is a randomized, double-blind, controlled and multi-center Phase III clinical trial to evaluate the safety and efficacy of ASC40 tablets combined with bevacizumab in the treatment of adult patients with recurrent glioblastoma. After standard radiotherapy and chemotherapy (temozolomide), the subject first experienced clinical recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, both male and female;
* 2. Histologically confirmed glioblastoma;
* 3. Patients with glioblastoma who have failed standard treatment (surgery, Stupp regimen), were diagnosed by MRI and evaluated by RANO standard to support the first recurrence. Stupp regimen needs to complete at least 6 medication cycles.

Exclusion Criteria:

* 1. Use low molecular weight heparin and warfarin within 35 days before randomization;
* 2. Arterial or venous thrombosis (such as cerebral infarction, myocardial infarction, venous thrombosis of lower limbs, arterial embolism of lower limbs, pulmonary embolism, etc.) occurred within 6 months before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  The time of progression or death from any cause in randomly grouped diseases (whichever comes first) was compared with the control group (evaluated by Independent Imaging Evaluation Committee [IRC])
Total survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  the time from random grouping to death, compared with the control group.

SECONDARY OUTCOMES:
Objective remission rate | Week 4 to Month 6 (every 8 weeks)
  It is evaluated once in the 4th week after using experimental drugs (experimental drug group or control group), and then every 8 weeks until the disease progresses or dies (evaluated by [IRC]).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital，Capital Medical University, Beijing, Beijing Municipality, China